CLINICAL TRIAL: NCT04942756
Title: GLYPALCARE STUDY - Multicenter, Randomized Study for Evaluating Continuous Glucose Monitoring (CGM) by Using FreeStyle Libre 2 (FSL2) for Preventing Hyperglycemia/Hypoglycemia Crisis in Advanced Oncological Patients With Known/Newly Diagnosed Type I/Type II Diabetes Mellitus (DM) in Palliative Care/ Supportive Care (PC/SC) Setting.
Brief Title: GLYPALCARE STUDY - Multicenter, Randomized Study for Evaluating Continuous Glucose Monitoring (CGM) by Using FreeStyle Libre 2 (FSL2) for Preventing Hyperglycemia/Hypoglycemia Crisis in Advanced Oncological Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Antea Foundation (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Antea-ARC-21-01
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Palliative Care; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes; Cancer; Terminal Cancer; Terminal Illness; End Stage Cancer; Advanced Cancer
Keywords: Palliative care; Diabetes; Cancer; Advanced cancer; End Stage Cancer; Terminal Cancer
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Mellitus; Neoplasms | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous Glucose Monitoring (Experimental): The FreeStyle Libre 2 Flash Glucose Monitoring System (FSL2) is a CGM device with real time alarms capability indicated for the management of diabetes in persons aged 4 and older. The Sensor holds eight (8) hours of data at a time. In order to have a daily diary of the Glucose level the patients or family or HCP must read the sensor (with reader or app) at least every height (8) hours. Every day at least three (3) scans of the sensor should be performed using the reader or the Smartphone App, generally at wake up in the morning, in the afternoon and at the time to go to sleep.
  The alarm system will be activated, so that the Glucose level is over the cut off limit of 180 mmol/L or when it is lower than the cut-off limit of 80 mmol/L, the patient and/or the family members and/or the caregiver will check the Glucose level by scanning the reader/smartphone over the sensor.
  Interventions: Device: Continuous Glucose Monitoring
- Standard Care (Active Comparator): This arm will perform the usual standard routine for blood glucose monitoring in patients with insulin therapy, that is represented by at least three finger pricks/die according to the usual standards routine of each center.
  Different frequency of finger pricks glucose measurements could be performed on the basis of health care professional patient assessment of each patient's needs.
  Interventions: Device: Standard Care

INTERVENTIONS:
Device: Continuous Glucose Monitoring — FSL2 is an integrated continuous glucose monitoring (CGM) system that provides continuous glucose measurements every minute to provide glucose levels, trends and alerts. It is composed by a sensor and a reader. The Sensor, to apply on the back of the arm, continuously measures glucose concentration in interstitial fluid and has an 8-hour memory capacity. The Sensor is factory calibrated, does not require finger stick calibration and can be worn for up to 14 days.
  The reader is a small handheld device that monitors glucose values in real-time to provide alerts and alarms which, when enabled, warn the user of Low Glucose, High Glucose or Signal Loss and prompt the user to scan the Sensor.
  The FSL 2 System is CE mark, it is commercially available and in the current study it is being used in accordance with approved labeling. No modifications of FSL2 System have been performed for the utilization in the current study.
  Arms: Continuous Glucose Monitoring
Device: Standard Care — The control group is represented by the usual standard way for blood glucose (BG) monitoring. The control group will use a lancing device for finger samples for collection of blood drop to be put in the test strips to be read in the Glucose meter. Lancing devices, lancets and test strips used in the comparison groups are CE marked and are used according to the user's instructions.
  Monitoring and/or self-monitoring of blood glucose using glucose meters and test strips provides quantitative measurements of fingerstick blood glucose at a single point in time for patients and their healthcare providers to monitor the effectiveness of glycemic control and make more immediate treatment with the right dosage of insulin. The usual standard routine for blood glucose monitoring in patients with DM and with insulin therapy is represented by at least three finger pricks/die according to the usual standards routine of each center.
  Arms: Standard Care

SUMMARY:
Cancer patients with known or newly diagnosed (i.e. iatrogenic) Diabetes Mellitus (DM) in Palliative/Supportive Care will be enrolled. Patients will be randomly assigned to one of two groups. Patients included in the first group will monitor glucose levels through Continuous Glucose Monitoring (CGM), using the FreeStyle Libre 2 (FSL2). The second group is represented by the usual standard way for blood glucose (BG) monitoring (lancing device for finger samples). An interim analysis is foreseen when the half of the expected events (hyperglycemic peaks) will be observed. In case the results of interim analysis show superiority of the CGM (FSL2) group patients of the second group will be switched.

DETAILED DESCRIPTION:
Diabete Mellitus (DM) represents an emerging factor with an impact on the severity and the management of symptoms (pain, dyspnoea, fatigue, nausea, vomiting, dehydration) in PC/SC patients leading to a reduced QoL of patients and family members. It has been noted that infrequent Blood Glucose (BG) monitoring might result in a not clear definition about whether symptoms are associated with the dying process or caused by diabetes, leading to inadequate symptoms management.

It is estimated that more than 30% of PC/SC patients can be affected by DM type I or type II. The incidence of diabetes seems to be six times greater in cancer patients than in the general population.

Despite this high incidence, implementation of standard Guidelines on monitoring BG levels in the PC/SC setting is lacking and the existing Guidelines are mainly based on expert experience rather than real data obtained from well design studies as evidenced by a recent review. Currently, the available tool used to evaluate BG in PC/SC patients is mainly represented by the punctual finger-samples procedure, which is usually performed only when there is a suspect of hyperglycemia/hypoglycemia or routinely in PC patients with known DM before meals administration. Punctual finger-samples procedure has many limitations: it is uncomfortable and painful for patients, it requires training to patients and family members by Health Care Providers (HCPs) and requires time to HPCs for preparing/conducting the procedures. As a consequence, BG monitoring in PC/SC patients (especially in home care settings) with known DM and newly diagnosed DM is very poorly and infrequently performed and represents a real unmet medical need.

Recently, a very innovative device, Freestyle Libre 2 (FSL2) (Abbott), has obtained a CE mark for Continuous Glucose Monitoring (CGM) in diabetic patients. The system includes a self-applied sensor with a size of two-stacked quarters, that is easy to apply on the back of the upper arm; it employs a pre-calibrated sensor that measures the tissue glucose concentration repeatedly for two weeks and has a duration of accuracy measurements of 14 consecutive days; interstitial Glucose levels are easily check with a painless one-second scan by a smartphone App or a Reader with results represented by latest glucose concentration and trend direction. The scan with the App or the Reader should be applied at least every 8 hours in order to have the recording of the glucose level. FSL2 has real-time glucose alarms that notify if glucose level is going too low or too high (Free Style Libre 2 User's Manual).

The rationale of the proposed study is based on the CGM system using FSL2, that is highly matching the need of Glucose level monitoring in PC/SC patients with known or newly diagnosed (i.e. iatrogenic) DM. FSL2 has no/very little discomfort for patients and it is not painful, it is easy to apply, it is not time-spending for family members and HCPs and it requires very brief training for patients and family members. The alarm system of FSL2 can aware patients, family members and HCPs at any moment when the glucose level is over a predefined cut off value, allowing to implement the appropriate interventions (i.e. insulin administration or insulin dose adjustment) in order to prevent and manage Symptomatic hyperglycemia crisis. The recent International Consensus on Recommendations on CGM data interpretation are showing that in particularly frail population, Glucose level are maintained for 50% of the time in a range between 70 mg/dL and 180 mg/dL and for 50% of the time in a range between 180 mg/dl and 250 mg/dl. According to that Recommendations, the alarm could be activated when glucose is over a cut off level of 180 mg/dL. The alarm activation allows patients themselves, family members, HCPs to provide patients with the most appropriate intervention (i.e. administration or adjustment of insulin dosage) in order to prevent glucose level reaching the peak of severe hyperglycemia (>250 mg/dl).

Similarly, FSL2 allows to monitor Glucose level decrease and to prevent severe hypoglycemic crisis (BG <50 mg/dL).

On this basis, we would like to evaluate CGM by using FSL2 as a tool for appropriately managing Glucose levels in PC/SC advanced oncological patients with known or newly diagnosed DM in order to prevent severe hypoglycemic/hyperglycemic crisis, in comparison to the current usual procedures (finger samples procedures).

CGM by using FSL2 could have a very positive impact in improving glucose level management in the PC/SC setting, especially in the home care setting, contributing to an improvement of the QoL of patients/family members and the HCPs attitude to the importance of glucose level monitoring. The results of this study could lead to a new standard of care in the management of patients with advanced cancer with a known/newly diagnosed DM in PC/SC settings.

The study is a multicenter, multinational, randomized, open label, parallel groups study, conducted in order to show superiority of CGM by using FSL2 in comparison to usual care procedures (finger samples) in reducing severe hyperglycemic peaks in PC/SC advanced oncological patients with known/newly diagnosed DM.

An interim analysis is foreseen when the half of the expected events (hyperglycemic peaks) will be observed. In case the results of interim analysis show superiority of the CGM (FSL2) group in respect to the control group, patients of the control group will be switched to CGM by using FSL2 and will be followed until the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged > or = 18 years
* Diagnosed with advanced oncological disease
* Known/newly diagnosed DM according to ADA criteria
* Need of a Insulin therapy and need of Glycemia Monitoring with at least three finger pricks/die
* Karnofsky Index >= 30
* Provision of signed and dated informed consent form

Exclusion criteria:

* Diagnosis of all types of Dementia
* Presence of severe psychiatric diseases/symptoms
* Kidney failure requiring dialysis
* Patients with implanted pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate CGM by using FSL2 in preventing severe hyperglycemia peaks | From recruitment until last followup (8 weeks)
  First severe hyperglycemic peak (>250 mg/dL) observed during evaluation

CONTACTS AND LOCATIONS:
Locations (6):
- Palliative care Service - Sheba Medical Centre, Ramat Gan, Israel
- Italy (4):
  - Antea Foundation, Roma
  - Centro di Cure Palliative "Insieme nella Cura" - Policlinico Universitario - Campus Bio-Medico (Roma), Roma
  - Unità Operativa Complessa di Oncologia Medica - Policlinico Univeristario Campus Bio-medico di Roma, Rome
  - Fondazione FARO, Torino
- Hospiz im Park, Arlesheim, Switzerland